CLINICAL TRIAL: NCT03651778
Title: Laboratory Analysis of Toxic Agents in Suspected GHB Poisoning, Clinical Course and Predictors of Hospitalization in GHB Poisoning, and Laboratory Analysis of Toxic Agents in Poisoning Induced by Others
Brief Title: GHB Poisoning and Poisoning Induced by Others
Status: Completed | Type: Observational
Sponsor: Odd Martin Vallersnes (Other)
Collaborators: Lovisenberg Diakonale Hospital (Other); Diakonhjemmet Hospital (Other); Oslo University Hospital (Other); University of Oslo (Other); Oslo Accident and Emergency Outpatient Clinic (Unknown)
Responsible Party: Sponsor-Investigator, Odd Martin Vallersnes, Professor, University of Oslo
Organization: University of Oslo (Other)
Other Study IDs: 2017/1880/REK
Record Dates: First submitted 2018-08-22; First posted 2018-08-29 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2023-11

CONDITIONS: Drug Toxicity
Keywords: GHB; gamma-Hydroxybutyric acid; Substances of abuse; Poisoning induced by others; Recreational drugs; Poisoning; Intoxication
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Poisoning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine, oral fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Suspected spiked drink exposure, no assault
- Suspected spiked drink exposure, sexual assault
- Suspected GHB exposure

SUMMARY:
Patients with suspected GHB poisoning presenting to Oslo Accident and Emergency Outpatient Clinic (Oslo Legevakt) or a hospital in Oslo (Oslo University Hospital Ullevål, Diakonhjemmet, Lovisenberg) will be included. Oral fluid and blood tests will be analyzed for recreational drugs. Clinical course will be charted, as well as treatment in the ambulance, emergency outpatient clinic and hospital to find predictors for when hospitalization is required.

In the second part of the study the investigators will analyze urine and blood samples from patients presenting to the Oslo Accident and Emergency Outpatient Clinic (Oslo Legevakt) with suspected substance poisoning induced by others, for toxic agents.

DETAILED DESCRIPTION:
Gammahydroxybutyrate (GHB) causes severe poisoning that requires emergency medical and hospital care. In addition, it is used as an anesthetic for planned sexual assault. Laboratory analyses will help assess whether today's clinical diagnostics of GHB poisoning are precise enough, possibly being a supplement to improve it. Can GHB poisoned patients be treated safely by emergency medical services or do these patients need hospitalization?

In case of substance poisoning induced by others, sampling could identify substances that are quickly excreted from the body. Today patients are referred to private laboratories the following day, delaying the diagnosis and missing short-term drugs.

Method: Prospective study. Oral fluid and blood samples will be collected from patients over 16 years of age where there is a clinical suspicion of GHB poisoning on arrival at Oslo Accident and Emergency Outpasient Clinic (Oslo Legevakt) or hospital (OUH Ullevål, Lovisenberg and Diakonhjemmet). Blood and urine samples will be collected from patients over the age of 16 who present at the Oslo Accident and Emergency Outpasient clinic (Oslo Legevakt) with suspected substance poisoning induced by others. In both pasient groups the investigators will also register age, gender, clinically suspected toxic agents, vital signs, clinical features and treatment.

The aims of this study are to see if the clinical diagnosis of GHB poisoning is precise enough, and whether more patients can be handled at an emergency outpatient level. Furthermore, analysis of blood and urine samples from patients who suspect they have been poisoned by substances induced by others, will be done to identify toxic agents.

ELIGIBILITY:
Inclusion Criteria:

Clinically suspected GHB poisoning means patients

* who are comatose or have varying level of consciousness,
* where there is absence of signs of opioid poisoning or poisoning with other agents,
* where there is no effect of naloxone,
* where there is information from a patient or companion about the intake of GHB
* or where there is a finding of GHB in the patient's belongings.

Exclusion Criteria:

* patients under 16 years of age

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to Oslo Accident and Emergency Outpatient Clinik (Oslo Legevakt) or Oslo hospitals with clinically suspected GHB poisoning.
  Patients presenting to Oslo Accident and Emergency Outpatient Clinic (Oslo Legevakt) with suspected substance poisoning induced by others within the last 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with confirmed GHB poisoning in blood or oral fluid samples, and what other drugs were detected. | Blood or oral fluid samples will be collected as soon as possible after presentation to the collaborating emergency health services, at the latest within 12 hours of presentation.
  Blood and oral fluid samples will be analyzed looking for GHB and the most commonly used recreational drugs (including ethanol).
Clinical factors at presentation predicting the necessity of hospital admission. | Clinical factors will be assessed at the initial presentation to emergency health services. Criteria for necessity of hospital admission will be assessed at 12 hours after presentation to hospital emergency department.
  We will do a multiple logistic regression analysis to identify factors associated with necessity of hospital admission. If during the clinical course of the poisoning episode the patient was intubated, had a GCS below 7, an arrhythmia requiring intervention, was admitted to an intensive care intake, or kept in hospital emergency department for more than 12 hours, the patient will be deemed as needing hospital admission as opposed to treatment in an emergency outpatient setting.
Recreational drugs (including ethanol) in blood and urine samples. | Blood and urine samples will be collected at presentation to emergency health services, if within 48 hours of the suspected ingestion.
  Blood and urine samples will be analyzed, looking for the most commonly used recreational drugs and for the drugs most often used in poisoning inflicted by others.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Institute of Health and Society, Oslo, Oslo County, Norway